CLINICAL TRIAL: NCT03475797
Title: Evaluation of Occipital Nerve Stimulation in Intractable Occipital Neuralgias: a Multicentric, Controlled, Randomized Study
Brief Title: Evaluation of Occipital Nerve Stimulation in Intractable Occipital Neuralgias
Acronym: StimO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision to stop the study prematurely due to insufficient inclusion.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC17_0013
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Occipital Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occipital Nerve Stimulation (ONS) (Experimental): Occipital nerve stimulation with percutaneous or surgical lead plus optimal medical management
  Interventions: Device: Occipital nerve stimulation; Other: Optimal Medical Management
- Optimal Medical Management (OMM) (Active Comparator): Optimal Medical Management according to what is done in routine clinical practice
  Interventions: Other: Optimal Medical Management

INTERVENTIONS:
Device: Occipital nerve stimulation — Occipital nerve stimulation with percutaneous or surgical lead
  Arms: Occipital Nerve Stimulation (ONS)
Other: Optimal Medical Management — Optimal Medical Management according to what is done in routine clinical practice : drug, psychobehavioral approach, acupuncture, sophrology, etc.

SUMMARY:
Medically intractable pain caused by occipital neuralgia can be very difficult to control with traditional pain management. Peripheral nerve stimulation which is used in migraines and cluster headache can be an alternative for these patients with occipital neuralgias when medical treatment and traditional pain management have failed (drugs for neuropathic pain, infiltrations, psychobehavioral approaches and multidisciplinary approach in a pain center). Occipital nerve stimulation consists to put a lead subcutaneously in front of the occipital nerve and to connect the lead to a pulse generator. A retrospective study of 60 patients was conducted in Nantes University Hospital. The results were good with the Visual Analog Scale (VAS) decreased from 8.4 preoperatively to 2.85 postoperatively. The medical quantification scale (MQS) was reduced to about 50% (18 preoperatively versus 9.9 postoperatively). Stimulation was quiet stable over time with a mean follow-up of 24 months (range 6 to 72 months). The aim of StimO is to confirm this result through a national controlled randomized multicenter study where occipital nerve stimulation will be compared to the optimal medical management.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 85 years old
* Chronic occipital neuralgias as defined by International Headache Society (IHS) more than 6 months with permanent pain associated or not with paroxysm
* Secondary occipital neuralgias (post-traumatic, post-surgery, major arthrosis, compression or lesion of the occipital nerve …)
* Chronic neuropathic pain according to the Neuropathic Pain Diagnostic Questionnaire (DN4 ≥ 4)
* Maximum pain on VAS ≥ 50/100
* Failure of medical treatment (association of neuropathic medication like antiepileptic and/or antidepressant and/or antalgic treatment like paracetamol, tramadol or morphine) and pain management in a pain Unit including multidisciplinary approach, physiotherapy, block test in C1-C2, radiofrequency rhizolysis, and/or corticosteroid infiltration of C2 according to the criteria defined by Health Authorities for spinal cord stimulation.
* Reduction of pain with Transcutaneous Electrical Nerve Stimulation (TENS) in occipital area
* Neurological examen has to be completed and must be normal except for the occipital neuralgia territory
* A negative pregnancy test for women with childbearing potential
* Women of childbearing potential must use appropriate method(s) of contraception during the clinical trial
* Patients must be capable of giving informed consent and must have signed informed consent
* Affiliation to an appropriate health insurance

Exclusion Criteria:

* Contraindication to the experimental medical devices
* Titanium related allergies
* Patients with contraindications to general anesthesia
* Complete anaesthesia in the C2/Great occipital nerve territory
* Drug or alcohol addiction
* Psychiatric disorders (psychiatric evaluation)
* Any medical or psychological problems which may interfere with a smooth conduction of the study protocol (e.g. cancer with a limited life expectancy)
* Need for intensive nursing care
* Difficulty in follow-up
* Pregnant or lactating women
* Women not using contraception
* Adults under a legal protection regime (guardianship, trusteeship, "sauvegarde de justice")
* Exclusion period for another study
* Simultaneous participation in another clinical trial except if that other trial does not affect the StimO study as approved and documented by the sponsor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of occipital nerve stimulation | 6 months
  Compare the decrease of pain (evaluated by visual analogic scale) after 6 months of treatment between the 2 groups (ONS / OMM)

SECONDARY OUTCOMES:
Decrease of medical treatment (i.e. decrease of Medication Quantification Scale (MQS) score) in the ONS group at 3 months | 3 months
  Evaluate the decrease of medical treatment (i.e. decrease of Medication Quantification Scale (MQS) score) after 3 months of occipital nerve stimulation in the ONS group
Decrease of medical treatment (i.e. decrease of Medication Quantification Scale (MQS) score) in the ONS group at 6 months | 6 months
  Evaluate the decrease of medical treatment (i.e. decrease of Medication Quantification Scale (MQS) score) after 6 months of occipital nerve stimulation in the ONS group
Maximum pain (using Visual Analogic Scale) | Up to 6 months
  Comparison of maximum pain (using Visual Analogic Scale) between the 2 groups (ONS/OMM)
Average pain (using Visual Analogic Scale) | Up to 6 months
  Comparison of average pain (using Visual Analogic Scale) between the 2 groups (ONS/OMM)
Relative decrease of pain (using Visual Analogic Scale) at 3 months | 3 months
  Comparison of the relative decrease of pain (using Visual Analogic Scale) at 3 months between the 2 groups (ONS/OMM)
Relative decrease of pain (using Visual Analogic Scale) at 6 months | 6 months
  Comparison of the relative decrease of pain (using Visual Analogic Scale) at 6 months between the 2 groups (ONS/OMM)
Efficacy of the treatment (using Migraine Disability Assessment (MIDAS) Test) at 3 months | 3 months
  Comparison of the efficacy of the treatment (using Migraine Disability Assessment (MIDAS) Test) at 3 months between the 2 groups (ONS/OMM)
Efficacy of the treatment (using Migraine Disability Assessment (MIDAS) Test) at 6 months | 6 months
  Comparison of the efficacy of the treatment (using Migraine Disability Assessment (MIDAS) Test) at 6 months between the 2 groups (ONS/OMM)
Quality of life (using EQ-5D-5L questionnaire) | Up to 6 months
  Comparison of the quality of life (using EQ-5D-5L questionnaire) between the 2 groups (ONS/OMM)
Quality of life (using Hamilton Anxiety and Depression (HAD) scale) | Up to 6 months
  Comparison of the quality of life (using Hamilton Anxiety and Depression (HAD) scale) between the 2 groups (ONS/OMM)

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - CHU Limoges, Limoges
  - Hôpital Pierre Wertheimer, Lyon
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - Hôpital Lariboisière, Paris
  - Hôpital Foch, Paris
  - CHU de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No